CLINICAL TRIAL: NCT04033302
Title: A Multi-Center Study of Multiple CAR T Cell Therapy for CD7-positive Hematological Malignancies
Brief Title: Multi-CAR T Cell Therapy Targeting CD7-positive Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-19005
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; T-cell Acute Lymphoblastic Lymphoma; Acute Myeloid Leukemia; NK Cell Lymphoma
Keywords: T-ALL; TCL; AML; NK lymphoma; CAR T; CD7
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Multiple CAR T cells to treat CD7-positive hematological malignancies
  Interventions: Biological: CD7-specific CAR gene-engineered T cells

INTERVENTIONS:
Biological: CD7-specific CAR gene-engineered T cells — Infusion of CD7-specific CAR-T cells

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of CAR T cell therapy against CD7-positive hematological malignancies using CD7 specific CAR T cells. The study also aims to learn more about the function of CD7 CAR T cells and their persistence in patients of hematological malignancies.

DETAILED DESCRIPTION:
Hematological malignancies including T-cell acute lymphoblastic leukemia (T-ALL), T cell lymphoma (TCL), natural killer cell lymphoma (NKL) and acute myeloid leukemia (AML) are aggressive diseases which may express the early T cell development molecule CD7.

T-ALL represents 15% of childhood and 25% of adult ALL, and T-ALL patients are prone to early disease relapse and suffer from poor outcomes. Several immunophenotypic classifications have been proposed. According to European Group for the Immunological Characterization of Leukemias (EGIL), the presence of cytoplasmic or membrane expression of CD3 defines T-ALL. Four subgroups are proposed: (TI) the immature subgroup or pro-T-ALL is defined by the expression of CD7 and cCD3; (TII) pre-T-ALL also expresses CD2 and/or CD5 and/or CD8; (TIII) or cortical T-ALL shows CD1a positivity; (TIV) finally, mature T-ALL is characterized by the presence of surface CD3 and CD1a negativity.

Over the past few years, T cells modified with lentiviral chimeric antigen receptor (CAR) gene have been studied in different clinical settings. CD7 is a T cell surface protein that plays important role in T cell-B cell interaction in early lymphoid development, displays membrane expression early during T cell development before TCR rearrangement, and persists through terminal stages of T cell development, and a well-known marker for T-ALL. CD7 is considered a promising target for the treatment of T-ALL, TCL, AML and NKL. In this study, we will investigate CD7 CAR-T in combination with alternative targeting CAR-T cells as a new strategy to treat hematological malignancies.

The T cells from patients or transplantation donors will be genetically modified with lentiviral CAR vector to recognize CD7 expressed on the surface of the cancer cells. The engineered T cells will be applied to patients through intravenous delivery.

The purpose of this clinical trial is to assess the feasibility, safety and efficacy of multiple CAR-T cell therapy in hematological malignancies. Another goal of the study is to learn more about the function of CAR T cells and their persistence in the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. Confirmed expression of CD7 or additional surface antigens in the cancer cells by immuno-histochemical staining or flow cytometry.
3. Karnofsky performance status (KPS) score is higher than 80 and life expectancy > 3 months.
4. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: cardiac ejection fraction ≥ 50%, oxygen saturation ≥ 90%, creatinine ≤ 2.5 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, total bilirubin ≤ 2.0mg/dL.
5. Hgb≥80g/L.
6. No cell separation contraindications.
7. Abilities to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
2. Active bacterial, fungal or viral infection not controlled by adequate treatment.
3. Known HIV or hepatitis C virus (HCV) infection.
4. Pregnant or nursing women may not participate.
5. Use of glucocorticoid for systemic therapy within one week prior to entering the trial.
6. Previous treatment with any gene therapy products.
7. Patients, in the opinion of investigators, may not be able to comply with the study.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion | a year
  Treatment-related adverse events are assessed by NCI CTCAE V4.0 criteria.

SECONDARY OUTCOMES:
Clinical response | a year
  Objective responses (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China